CLINICAL TRIAL: NCT03721250
Title: Comparison of Thoracic Epidural Analgesia and Intercostal Blockade in Patients Undergoing Thoracotomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Associated professor, Ankara University
Other Study IDs: Ank230918
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Analgesia, Postoperative
MeSH Terms: conditions — Agnosia | interventions — Injections, Epidural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thoracic epidural: patients receiving thoracic epidural
  Interventions: Other: epidural

INTERVENTIONS:
Other: epidural — thoracic epidural analgesia

SUMMARY:
Postoperative pain is an important issue after thoracotomy operations. Thoracic epidural analgesia is most popular analgesic method, but sometimes it is not sufficient for pain. This study is designed to compare intercostal block with thoracic epidural analgesia in patients undergoing thoracotomy

ELIGIBILITY:
Inclusion Criteria:

lung cancer

Exclusion Criteria:

patient refusal bleeding diathesisi emergency cases

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thoracotomy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
verbal analog score | postoperative 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided